CLINICAL TRIAL: NCT03764384
Title: An Observational Study in People With Amyotrophic Lateral Sclerosis to Validate Tidal /End-Tidal CO2, Measured by the N-Tidal C™ Against Directly Measured PaCO2 and to Determine the Ease of Home Use of the Device
Brief Title: Validation Of Tidal/End -Tidal CO2 in ALS
Acronym: VOTECO2ALS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: Motor Neurone Disease Association (Unknown); Innovate UK (Other Government); DOCATEF (Unknown); TidalSense (Industry)
Responsible Party: Sponsor
Other Study IDs: P02366
Record Dates: First submitted 2018-08-29; First posted 2018-12-05 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Motor Neuron Disease; Amyotrophic Lateral Sclerosis
Keywords: PaCO2; N-Tidal C Device; Self-monitoring; CO2 waveforms
MeSH Terms: conditions — Motor Neuron Disease; Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hospital Monitoring Group - ALSFRS-R cohort: All patients will be first recruited to this cohort unless at their first visit the investigator deems them eligible for the Home Monitoring Device Group. At the initial screening visit, all patients recruited into the study will undergo routine assessments according to the existing MND protocol, and additionally complete the ALSFRS-R symptom-based assessment questionnaire by interview with the study researchers (with assistance from spouse, family member or carer if required). Patients will continue to complete the ALSFRS-R symptom-based questionnaire at each clinic attendance.
- Home Monitoring Cohort: If eligible patients will use the N Tidal CTM, up to 3 times a day (morning, midday and evening) throughout the home monitoring period until the final outpatient clinic visit.
  In addition subjects will complete a weekly diary symptom monitoring diary which asks them about their respiratory symptoms, GP attendances, respiratory infections. Patients routine standard of care assessments will also be documented according to the protocol as well as completing the ALSFRS-R at each visit.

SUMMARY:
The study team propose that a new, hand-held test device may be valuable in the management of breathing failure in patients with Motor Neurone Disease (MND). The study team need to validate this device against the current gold standard of blood gas analysis and determine whether people with MND can use it at home. The new device, called 'N-Tidal C™' measures the carbon dioxide (CO2) in expired breath. At the end of the breath (end tidal) the CO2 level gives an indication of the CO2 in the person's arterial blood. Ventilatory failure is diagnosed at present using the value of CO2 in the arterial blood, but usually this can only be measured in specialist clinics. The study will determine if the end tidal CO2 measured by the new device agrees with CO2 measured on a blood test in clinic and also whether or not the device is practical for home use. The team will analyse the output of the device during home monitoring to see if changes in the pattern of CO2 in the expired breath identify, or even predict, the development of breathing failure in the community. With the results of these measures and detailed information about the patients in Papworth's clinic, recruited to this study, collected over a year the team will design a follow on study to see if using the new device at home can improve survival and quality of life for people with MND.

DETAILED DESCRIPTION:
This is a prospective, observational study of patients attending Royal Papworth Hospital's weekly MND clinic. If a patient decides to participate in the study, they will continue to receive all normal care. Researchers will ask permission to review the results of any medical investigations and tests previously undertaken, by looking in medical records and will collect new data prospectively. There will be two groups of patients recruited:

A).Hospital Questionnaire Monitoring Group (12 months) for up to 200 patients who will:

i) Have four routine hospital based assessments (every 3 months, standard care) ii) Above usual care: completion of the ALSFRS-R questionnaire at each clinic (4 in total. The ALSFRS-R (Amyotrophic Lateral Sclerosis Functional Rating Score-Revised) measures range of difficulties that people with MND can have in their daily lives. The results from this questionnaire help to measure the severity of MND symptoms, and how fast the disease is progressing. B). Home Device Monitoring Group (12-24 months) for 30 patients These participants patient will be given a portable monitoring device (called the N-Tidal C) to record their breathing pattern in clinic and at home and have: i) Four to six routine hospital based assessments (every 3 months, standard care). At the discretion of the investigator this may be at each clinic visit up to a total of 24 months ii) Completion of an ALSFRS-R symptom questionnaire at each visit (4-6 in total). At the discretion of the investigator this may be at each clinic visit up to a total of 24 months iii) Telephone consultation 2 weeks after commencing home monitoring to validate correct and safe use of the device (1 in total) iv) Completion of a supervised N-Tidal C breath record at each clinic visit (4 to 6 total). At the discretion of the investigator this may be at each clinic visit up to a total of 24 months v) Completion of a weekly symptom diary (up to 52 in total). At the discretion of the investigator this may continue up to 24 months vi) Home monitoring with N-Tidal C for 75 seconds, up to 3 times per day (up to study finish). SA 02 introduced an additional modified breath holding manoeuvre for home monitoring patients in clinic.

The range of 4 to 6 assessments covers the eventuality that participants may start in group A and transfer to group B as their condition changes. This will be determined by the treating doctor and will be based upon their lung function, limb weakness and whether they (or a carer) are able to use the device. During the home monitoring trial, data collected by the N-Tidal C device will be downloaded at each clinic visit, to check that the device is correctly recording data. Researchers will not be able to analyse the data collected by the device.

Only the information obtained from the standard measurements (standard care) will be used to decide when a patient needs help with their breathing at night time by starting a ventilator. A patient participating in the Home Monitoring Group will continue to use their N-Tidal C device to record their daytime breathing up to 3 times per day, after they start using a ventilator.

ELIGIBILITY:
Inclusion Criteria:

- 1. Male or female with a diagnosis of definite or probable Motor Neurone Disease according to El Escorial criteria.

2. Willing and able to provide informed consent.

Exclusion Criteria:

1. Lung, chest wall, neuromuscular, cardiac or other comorbidity or abnormality that would markedly affect spirometry and/or other measures of lung function or TBCO2 measurements. To be judged by the CI.
2. Tracheostomy in situ

Additional Eligibility Criteria for Home Monitoring patients Patients invited to use the N-Tidal CTM data collecting device within the study would be selected using the following additional inclusion criteria. These patients in theory would be most likely to get reliable results from the capnometer, be candidates for NIV, and to reach one of the study end-points within the follow-up period.

Home monitoring Inclusion Criteria:

1. Not in ventilatory failure at the start of the study (PaCO2 < 6.0 KPa)
2. Sufficient manual dexterity and arm strength to use the device (or have a live-in carer/spouse/family member able to assist and willing to do so).
3. Verified able to use the device (by trial with dummy device).
4. Stated intention at the start of the study that they will accept NIV if they develop ventilatory failure.

Home Monitoring Exclusion Criteria

1. In the opinion of the clinical investigator, the participant would have difficulty completing the study procedures consistently.
2. Established on NIV treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will have previously been diagnosed with Motor Neurone Disease by a neurologist. Study participants will be recruited from patients attending weekly Motor Neurone Disease clinics within the RSSC at Royal Papworth Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-06-04 (Estimated); Study Completion 2021-06-04 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of interest is the degree of agreement between end tidal CO2 measured by the N-Tidal CTM device and PaCO2 from arterial blood gas analysis. | At each clinic visit through to study completion up to 24 months
  Arterial blood gas (measured in kPa) will be compared to the end tidal CO2 (kPa) measured from the N-Tidal CTM device. The measurements will be taken within 20 minutes of each other. The paired CO2 measures from N-Tidal CTM device and from ABG will be assessed for agreement. The results will be displayed graphically using a Bland Altman Plot and the mean difference, the standard deviation of the mean difference and confidence intervals for 95% limits of agreement will be reported.

SECONDARY OUTCOMES:
Identify when an MND patient requires additional support with their breathing, in the form of starting NIV as derived from the CO2 measurement (kPA) and Respiratory Rate (RR) per minute from the N-Tidal CTM device. | At each clinic visit through to study completion up to 24 months
  The waveforms taken from the N-Tidal CTM device will be analysed to give an end tidal CO2 (kPa) value and the mean and standard deviation of Respiratory rate per minute. Assuming there is an acceptable level of agreement between the two methods of measuring CO2 the data will be reviewed to establish if the end tidal measurement identified the onset of ventilatory failure before the clinic visit where it was confirmed on an arterial blood gas. After inspection of the data a judgement will be made on whether the correct measure is an individual result >6kPa or whether 2 or more consecutive measures >6 kPa would be the most reliable measure to conclude that ventilatory failure has now developed. For those participants who develop a PaCO2 > 6 kPa, the amount of time by which this predates the confirmatory blood gas will be reported in weeks.
Identify when an MND patient develops a treatable respiratory condition, such as an infection as derived from the CO2 measurement (kPA) and Respiratory Rate (RR) per minute from the N-Tidal CTM device.. | At each clinic visit through to study completion up to 24 months
  The mean end tidal CO2 (kPa) and the mean RR taken from the N-Tidal CTM device on the day before and the day of an identified respiratory event (from the symptom diary) will be examined to see if there is a reproducible change in the signal that might indicate that a respiratory event has occurred assuming in the future that the device will be monitored remotely.

OTHER OUTCOMES:
Any adverse events (AEs) reported during performing the study procedures | At each clinic visit through to study completion up to 24 months
  Safety outcome
Any adverse device events (ADEs | At each clinic visit through to study completion up to 24 months
  Safety outcome
Visual analogue scale (VAS) to record 'ease of use' of the N-Tidal C™ device during the study and at study completion | At each clinic visit through to study completion up to 24 months
  Patient outcome measure. VOTECO2ALS 'Ease of use Questionnaire' has been devised by the study team to gather patient feedback on their participation in the trial and how they have found using the device. The scale has a series of statements and patients are asked to choose one of the following 5 options; disagree strongly, disagree, neither agree or disagree, agree, agree strongly. A 'disagree' response would represent a poor outcome in regards to the study design and device use where as an 'agree' option would be a better outcome in regards to the study design and usability of the device. The feedback from the subjects on ease of use will be examined for common themes.

CONTACTS AND LOCATIONS:
Overall Officials: Ian E Smith, MA MD F.R.C.P, Principal Investigator — Royal Papworth NHS Hospital
Locations (1):
- Royal Papworth NHS Foundation Trust, Papworth Everard, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bourke SC, Tomlinson M, Williams TL, Bullock RE, Shaw PJ, Gibson GJ. Effects of non-invasive ventilation on survival and quality of life in patients with amyotrophic lateral sclerosis: a randomised controlled trial. Lancet Neurol. 2006 Feb;5(2):140-7. doi: 10.1016/S1474-4422(05)70326-4. PMID 16426990
- [Background] COPD clinical trial : NIHRCRN 19599, ISRCTN 56492264
- [Background] O'Neill CL, Williams TL, Peel ET, McDermott CJ, Shaw PJ, Gibson GJ, Bourke SC. Non-invasive ventilation in motor neuron disease: an update of current UK practice. J Neurol Neurosurg Psychiatry. 2012 Apr;83(4):371-6. doi: 10.1136/jnnp-2011-300480. Epub 2011 Aug 17. PMID 21849339
- [Background] Checketts MR, Alladi R, Ferguson K, Gemmell L, Handy JM, Klein AA, Love NJ, Misra U, Morris C, Nathanson MH, Rodney GE, Verma R, Pandit JJ; Association of Anaesthetists of Great Britain and Ireland. Recommendations for standards of monitoring during anaesthesia and recovery 2015: Association of Anaesthetists of Great Britain and Ireland. Anaesthesia. 2016 Jan;71(1):85-93. doi: 10.1111/anae.13316. Epub 2015 Nov 19. PMID 26582586
- [Background] Banerjee SK, Davies M, Sharples L, Smith I. The role of facemask spirometry in motor neuron disease. Thorax. 2013 Apr;68(4):385-6. doi: 10.1136/thoraxjnl-2012-201804. Epub 2012 Jul 27. No abstract available. PMID 22843559
- See also: NICE guideline NG42: MND assessment and management — http://www.nice.org.uk/guidance/ng42/chapter/Recommendations
- See also: 4. NICE Technology Appraisal Guidance TA20 : Guidance on the use of Riluzole (Rilutek) for the treatment of Motor Neurone Disease — http://www.nice.org.uk/guidance/ta20